CLINICAL TRIAL: NCT04910568
Title: An Open-Label, Multicenter, Phase Ib Trial Evaluating the Safety, Pharmacokinetics, and Activity of Cevostamab as Monotherapy and Cevostamab Plus Pomalidomide and Dexamethasone or Cevostamab Plus Daratumumab and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study Evaluating the Safety, Pharmacokinetics, and Activity of Cevostamab in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: CAMMA 1
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO42552; 2021-000238-33 (EudraCT Number)
Record Dates: First submitted 2021-05-27; First posted 2021-06-02 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — tocilizumab; pomalidomide; daratumumab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single-Agent Cevostamab (Arm A) (Experimental): Cohort A1S is a safety run-in arm evaluating cevostamab administered in 28-day cycles on a modified weekly schedule.
  Cohort A1E, an expansion cohort, has been opened and finished enrolling participants. Participants will be treated with single-agent cevostamab administered in 28-day cycles on a modified weekly schedule.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab; Drug: Dexamethasone
- Cevostamab plus Pomalidomide and Dexamethasone (Pd) (Arm B) (Experimental): Participants will be treated with cevostamab monotherapy during a 14-day period prior to the start of pomalidomide treatment (cevostamab pre-phase).
  Cohort B1S is a safety run-in arm evaluating cevostamab and Pd administered in 28-day cycles every 2 weeks (Q2W) followed by every 4 weeks (Q4W) schedule. Additional safety run-in cohort(s) with lower target dose levels of cevostamab may be opened prior to opening the expansion cohorts.
  Two target dose levels of target dose level 1 (DL1) and lower dose level -1 (DL-1) of cevostamab will be selected for randomization in expansion cohorts. Expansion cohorts will follow the same Q2W/Q4W dosing schedule as Cohort B1S.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab; Drug: Pomalidomide; Drug: Dexamethasone
- Cevostamab plus Daratumumab and Dexamethasone (Dd) (Arm C) (Experimental): Cohort C1S is a safety run-in arm evaluating cevostamab and Dd administered in 21 day cycles from Cycle(C)1 - C8 every 3 weeks (Q3W) and 28-day cycles from C9 onwards Q4W. Additional safety run-in cohort(s) with lower target dose levels of cevostamab may be opened prior to opening the expansion cohorts.
  Two target dose levels of DL1 and DL-1 of cevostamab will be selected for randomization in expansion cohorts. Expansion cohorts will follow the same Q3W/Q4W dosing schedule as Cohort C1S.
  Interventions: Drug: Cevostamab; Drug: Tocilizumab; Drug: Daratumumab; Drug: Dexamethasone

INTERVENTIONS:
Drug: Cevostamab — Cevostamab will be administered intravenously on a 28-day cycle, up to a total of 13 cycles (Arm A), in 28-day cycles Q2W followed by Q4W (Arm B) and in 21 day cycles from C1-C8 Q3W and 28-day cycles from C9 onwards Q4W (Arm C). For Arm A, participants have the option to enter re-treatment after Cycle 13. For Arms B and C, participants can be treated until disease progression or unacceptable toxicity.
Drug: Tocilizumab — Tocilizumab will be administered for the treatment of cytokine release syndrome (CRS) when necessary.
  Other Names: Actemra/RoActemra
Drug: Pomalidomide — Pomalidomide will be administered orally (PO) on a 28-day cycle.
  Arms: Cevostamab plus Pomalidomide and Dexamethasone (Pd) (Arm B)
Drug: Daratumumab — Daratumumab will be administered subcutaneously (SC) on 21 day (C1-8) and 28-day cycles (C9 onwards).
  Arms: Cevostamab plus Daratumumab and Dexamethasone (Dd) (Arm C)
Drug: Dexamethasone — Arm A: Dexamethasone will be administered as a premedication.
  Arms B and C: Dexamethasone will be administered via IV or orally at 20 mg as study investigational medicinal product.

SUMMARY:
This Phase Ib, multicenter, open-label study will evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of cevostamab monotherapy, cevostamab plus pomalidomide and dexamethasone (Pd) or cevostamab plus daratumumab and dexamethasone (Dd) which will be administered to participants with relapsed or refractory multiple myeloma (R/R MM) via intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* Life expectancy of at least 12 weeks
* Agreement to provide bone marrow biopsy and aspirate samples
* Resolution of adverse events from prior anti-cancer therapy to Grade <=1
* Measurable disease
* For women of childbearing potential: agreement to remain abstinent or use contraception, during the treatment period (including treatment interruptions) and for at least 5 months after the last dose of cevostamab and at least 3 months after the last dose of tocilizumab was administered
* For men: agreement to remain abstinent or use a condom, and agreement to refrain from donating sperm, during the treatment period, and for at least 2 months after the last dose of tocilizumab was administered to avoid exposing the embryo and sexual partner Additional Arm A-Specific Inclusion Criteria
* Diagnosis of R/R MM for which no established therapy for MM is appropriate and available, or intolerance to those established therapies Additional Arm B-Specific Inclusion Criteria
* For Cohort B1S: Participants with R/R MM who have received at least two prior lines of treatment
* For Cohort B2S and additional cohorts: Participants with R/R MM who have received at least 1 prior line of treatment
* Agreement to comply with all requirements of the pomalidomide pregnancy prevention program
* For women of childbearing potential: agreement to remain abstinent or use two reliable methods of contraception starting at least 4 weeks prior to, during the treatment period, and for at least 4 weeks after the last dose of pomalidomide was administered
* For men: agreement to remain abstinent or use a condom during the treatment period and for at least 4 weeks after the last dose of pomalidomide, (even if he has undergone a successful vasectomy) and agreement to refrain from donating sperm and blood during this same period Additional Arm C-Specific Inclusion Criteria
* For Cohort C1S: Participants with R/R MM who have received at least two prior lines of treatment
* For Cohort C2S and additional cohorts: Participants with R/R MM who have received at least 1 prior line of therapy
* For women of childbearing potential: agreement to remain abstinent or use contraceptive methods during the treatment period and for at least 102 days after the last dose of daratumumab was administered
* For men: agreement to remain abstinent or use a condom during the treatment period and for at least 102 days after the last dose of daratumumab was administered to avoid exposing the embryo, and agreement to refrain from donating sperm during this same period

Exclusion Criteria:

* Prior treatment with cevostamab or another agent targeting FcRH5
* Inability to comply with protocol-mandated hospitalization and activities restrictions
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 5 months after the last dose of cevostamab or within 3 months after the last dose of tocilizumab (if applicable).
* Prior use of any monoclonal antibody, radioimmunoconjugate, or antibody-drugconjugate as anti-cancer therapy within 4 weeks before first study treatment, except for the use of non-myeloma therapy
* Prior treatment with systemic immunotherapeutic agents, including, but not limited to, cytokine therapy and anti-CTLA4, anti-PD-1, and antiPD-L1 therapeutic antibodies within 12 weeks or 5 half-lives of the drug, whichever is shorter, before first study treatment
* Prior treatment with chimeric antigen receptor T (CAR T)-cell therapy within 12 weeks before first study treatment
* Treatment with radiotherapy within 4 weeks (systemic radiation) or 14 days (focal radiation) prior to first study treatment
* Treatment with any chemotherapeutic agent or other anti-cancer agent (investigational or otherwise) within 4 weeks or 5 half-lives of the drug, whichever is shorter, prior to first study treatment
* Autologous SCT within 100 days prior to first study treatment
* Prior allogeneic stem cell transplant(ation) (SCT)
* Circulating plasma cell count exceeding 500/micro L or 5% of the peripheral blood white cells
* Prior solid organ transplantation
* History of autoimmune disease
* History of confirmed progressive multifocal leukoencephalopathy
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Known history of amyloidosis
* Lesions in proximity of vital organs that may develop sudden decompensation/deterioration in the setting of a tumor flare
* History of other malignancy within 2 years prior to screening
* Known treatment-related, immune-mediated adverse events associated with prior checkpoint inhibitors
* Current or past history of central nervous system (CNS) disease, such as stroke, epilepsy, CNS vasculitis, neurodegenerative disease, or CNS involvement by MM
* Significant cardiovascular disease
* Symptomatic active pulmonary disease or requiring supplemental oxygen
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection
* Known or suspected chronic active Epstein-Barr virus (EBV) infection
* Recent major surgery within 4 weeks prior to first study treatment
* Positive serologic or PCR test results for acute or chronic hepatitis B virus (HBV) infection
* Acute or chronic hepatitis C virus (HCV) infection
* Known history of Grade >= 3 CRS or immune effector cell-associated neurotoxicity syndrome (ICANS) with prior bispecific therapies
* Known history of hemophagocytic lymphohistiocytosis (HLH) or macrophage activation syndrome (MAS)
* Active symptomatic coronavirus disease 2019 (COVID-19) infection at study enrollment or requiring treatment with intravenous (IV) antiviral where the last dose of IV antiviral treatment was given within 14 days prior to first study treatment. Patients with active COVID-19 infection must have clinical recovery and two negative antigen tests at least 24 hours apart prior to first study treatment
* Positive and quantifiable EBV polymerase chain reaction (PCR) or Cytomegalovirus (CMV) PCR prior to first study treatment
* Known history of HIV seropositivity
* Administration of a live, attenuated vaccine within 4 weeks before first study treatment or anticipation that such a live attenuated vaccine will be required during the study
* Treatment with systemic immunosuppressive medications, with the exception of corticosteroid treatment <=10 mg/day prednisone or equivalent, within 2 weeks prior to first study treatment
* History of illicit drug or alcohol abuse within 12 months prior to screening, in the investigator's judgment Additional Arm B-Specific Exclusion Criteria
* Pregnant or breastfeeding, or intending to become pregnant 4 weeks prior to initiation of study treatment, during the study, (including treatment interruptions) or within 4 weeks after the last dose of pomalidomide
* Significant cardiovascular disease (such as, but not limited to, New York Heart Association Class III or IV cardiac disease, myocardial infarction within the last 12 months, uncontrolled arrhythmias, or unstable angina)
* History of erythema multiforme, Grade >=3 rash, blistering, or severe hypersensitivity to prior treatment with immunomodulatory drugs such as thalidomide, lenalidomide, or pomalidomide
* Inability to tolerate thromboprophylaxis, or contraindication to thromboprophylaxis
* GI disease that might significantly alter absorption of oral drugs Additional Arm C-Specific Exclusion Criteria
* Pregnant or breastfeeding, or intending to become pregnant during the study or within 102 days after the last dose of daratumumab
* Known hypersensitivity to biopharmaceuticals produced in CHO cells or any component of daratumumab formulations
* Known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) <50% of predicted normal
* Known moderate or severe persistent asthma within the past 2 years, or current uncontrolled asthma of any classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2029-12-10 (Estimated); Study Completion 2029-12-10 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose (RP2D) | Baseline up to approximately 4 years
Percentage of Participants with Adverse Events | Baseline up to approximately 4 years
Percentage of Dose Interruptions | Baseline up to approximately 4 years
Percentage of Dose Reductions | Baseline up to approximately 4 years
Percentage of Dose Intensity | Baseline up to approximately 4 years
Percentage of Treatment Discontinuation | Baseline up to approximately 4 years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Baseline up to approximately 4 years
Complete Response/Stringent Complete Response (CR/sCR) Rate | Baseline up to approximately 4 years
Rate of Very Good Partial Response (VGPR) or Better | Baseline up to approximately 4 years
Progression-free Survival (PFS) | Start of study treatment to first date of disease progression or death from any cause, whichever occurs first (up to approximately 4 years)
Duration of Response (DOR) | From first partial response (PR) or better until the first date of disease progression or death from any cause, whichever occurs first (up to approximately 4 years)
Time to First Response (for Participants who Achieve a Response of Partial Response (PR) or Better) | Baseline up to approximately 4 years
Time to Best Response (for Participants who Achieve a Response of PR or Better) | Baseline up to approximately 4 years
Minimal Residual Disease (MRD) Negativity | Baseline up to approximately 4 years
Overall Survival (OS) | Baseline up until death from any cause (up to approximately 4 years)
Serum Concentration of Cevostamab at Specified Timepoints | Cevostamab Pre-Phase (CPP) Day (D) 1 up to approximately 3 years
Total Exposure (Area Under the Concentration-time Curve [AUC]) of Cevostamab | CPP D1 up to approximately 4 years
Maximum Observed Serum Concentration (Cmax) of Cevostamab | CPP D1 up to approximately 4 years
Minimum Observed Serum Concentration (Cmin) of Cevostamab | CPP D1 up to approximately 4 years
Clearance of Cevostamab | CPP D1 up to approximately 4 years
Volume of Distribution at Steady State of Cevostamab | CPP D1 up to approximately 4 years
Number of Anti-drug Antibody (ADAs) Against Cevostamab at Baseline | Baseline
Percentage of Participants with ADAs Against Cevostamab During the Study | Up to approximately 4 years
Serum Concentration of Pomalidomide | From Cycle 1 Day 1 through Cycle 6 Day 15. Each cycle=28 days
Serum Concentration of Daratumumab | From C1D1 until disease progression or unexpected toxicity. Cycles 1-8 are 21 days and Cycle 9 onward are 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (27):
- United States (5):
  - City of Hope, Duarte, California
  - City of Hope - Lennar Foundation Cancer Center, Irvine, California
  - Colorado Blood Cancer Institute (CBCI) at Presbyterian/ St. Luke's Medical Center, Denver, Colorado
  - Karmanos Cancer Institute., Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
- Australia (2):
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network, Toronto, Ontario
- Fakultni Nemocnice Ostrava, Ostrava, Czechia
- Rigshospitalet, København Ø, Denmark
- France (2):
  - Hôpital Saint-Louis, Paris
  - CHU de Poitiers - La Miletrie, Poitiers
- Rambam Medical Center, Haifa, Israel
- Italy (2):
  - Asst Papa Giovanni Xxiii, Bergamo, Lombardy
  - A.O. Spedali Civili Di Brescia-P.O. Spedali Civili, Brescia, Lombardy
- Yamagata University Hospital, Yamagata, Japan
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Pratia Onkologia Katowice, Katowice
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Późna
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No